CLINICAL TRIAL: NCT07025590
Title: Effect of Exercise on Tapering Antipsychotics in Patients With Psycho-cardiological Disease: a Multicenter, Randomized Controlled, Non-inferior Clinical Study
Brief Title: Effect of Exercise on Tapering Antipsychotics in Patients With Psycho-cardiological Disease(EXTRA-study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Huan Ma, Deputy Director of Cardiology, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-198-01
Record Dates: First submitted 2025-04-15; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases (CVD); Depression Anxiety Disorder
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Escitalopram; Fluoxetine; Duloxetine Hydrochloride; Paroxetine; Venlafaxine Hydrochloride; Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise and medicine (Active Comparator): Exercise:Moderate-intensity continuous movement(MICT) The drugs include: sertraline, escitalopram, fluoxetine, duloxetine, paroxetine, venlafaxine, and fluvoxamine
  Interventions: Behavioral: Moderate-intensity continuous movement and Antipsychotics intervention
- medicine (Active Comparator): The drugs include: sertraline, escitalopram, fluoxetine, duloxetine, paroxetine, venlafaxine, and fluvoxamine
  Interventions: Drug: Antipsychotics intervention(sertraline, escitalopram, fluoxetine, duloxetine, paroxetine, venlafaxine, and fluvoxamine)

INTERVENTIONS:
Behavioral: Moderate-intensity continuous movement and Antipsychotics intervention — On the basis of Antipsychotics intervention, Patients in the exercise group should start exercise intervention as soon as possible after completing baseline examination, and need to complete a training plan of at least 36 times, 3 times/week. At the beginning of each training session, patients need to warm up for 5-10 minutes, mainly jogging and stretching exercises. After the warm-up, the patient enters the training phase, the heart rate reserve is 70% to 85%, and after the training, the patient performs 10-15 minutes of recovery exercise, mainly jogging, slow walking and stretching. The specific exercise plan is formulated according to the patients' own aerobic capacity assessment, and the principle of formulation is gradual and individual. At each training session, patients were asked about their perceived fatigue level to adjust the training intensity.
  Arms: Exercise and medicine
Drug: Antipsychotics intervention(sertraline, escitalopram, fluoxetine, duloxetine, paroxetine, venlafaxine, and fluvoxamine) — Patients maintained regular medication during the intervention period, and returned to the doctor every two weeks, and the psychiatrist decided whether to maintain the current dose or gradually reduce the dose based on the patient's symptoms and diagnosis. Psychiatrists, unaware of patient groupings, use supportive measures to help manage adverse reactions.
  Arms: medicine

SUMMARY:
Psycho-Cardiological Disease studies the complex links between the cardiovascular system and emotions. The two diseases are now the focus of public health organizations, forming a vicious circle of mutual influence. Anxiety and depressive symptoms are three to four times more common in patients with cardiovascular disease than in the general population, and about 15 to 18 percent of patients with coronary heart disease also have major depression, while 25 to 30 percent show significant depressive symptoms. At least 20% of patients with chronic heart failure have some degree of depression. In addition, the probability of cardiovascular events is 2.5 times higher in patients with two hearts, the risk of recurrence of cardiovascular events is heightened, and is strongly associated with higher mortality. At present, the common treatment methods show different advantages and disadvantages, for example, Antipsychotics treatment is a common means of depression/anxiety symptoms, with rapid onset, significant efficacy, wide application and other advantages. However, medications often struggle to fully relieve symptoms, have a high recurrence rate, and can have side effects. Psychotherapy as a traditional intervention method for mental disorders. Its advantages are long-lasting efficacy and no Antipsychotics dependence, but the effect is slower, and patients need to invest more time, energy and financial resources, and the psychological burden is also heavier. In recent years, exercise therapy, as a safe intervention without significant side effects, has been gradually included in a number of international clinical guidelines, and is regarded as the first-line recommended treatment for mild to moderate depression. Research has shown that exercise can effectively relieve anxiety and depression symptoms through a variety of mechanisms, such as lowering cortisol levels, regulating autonomic nervous system function, and reducing stress responses. A study of aerobic exercise in patients with Psycho-Cardiological Disease showed that a 16-week exercise intervention significantly reduced patients' depression scores and significantly improved mood and cognitive function. In addition, it has been validated in multiple studies that exercise can significantly reduce anxiety and depression symptoms by enhancing neuroplasticity, promoting neurogenesis and synaptic remodeling, improving cognitive and emotional regulation. These findings provide a strong theoretical and practical basis for the application of exercise therapy in the comprehensive management of Psycho-Cardiological Disease. The above studies provide important theoretical support for the treatment of biheart disease with exercise, but most studies focus on scale scores, biomarkers, and changes in social behavior. It is well known that antidepressant or anti-anxiety drugs can have many side effects due to their dosage, duration and long-term use, which in turn poses a potential risk to the overall health and quality of life of patients. Therefore, it is of significant clinical significance and research value to explore whether exercise as an adjunct therapy can effectively reduce the use of Antipsychotics and shorten the withdrawal period. This will not only help optimize personalized treatment plans, provide scientific basis for clinical decision-making, but also promote the development of Psycho-Cardiological Disease treatment to the direction of precision and integration.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with depression/anxiety;
2. Continued use of SSris and SNris for six months prior to study start;
3. Aged between 18 and 70;
4. Confirmed cardiovascular disease (such as chronic stable coronary heart disease, heart failure, cardiomyopathy, arrhythmia, valvular heart disease, cardiac surgery, cardiac intervention, ischemia with non-obstructive coronary artery disease, etc.);
5. The patients voluntarily participated in the study, signed a written informed consent, and were willing to cooperate with the follow-up.

Exclusion Criteria:

1. currently has mania or hypomania, or a history of bipolar disorder and any mental disorders (current and previous);
2. organic brain injury, etc., or serious non-cardiovascular system diseases (such as advanced cancer);
3. Unable to participate in sports training or have drug contraindications;
4. Current alcohol, drug abuse, drug use or suicidal intent;
5. Patients who were receiving other doses of eligible drugs and other antidepressants were excluded from the trial;
6. Myocardial infarction <2 weeks or unstable angina attack period;
7. Severe and uncontrolled arrhythmia;
8. Acute heart failure stage;
9. Severe and symptomatic obstruction of the outflow tract;
10. Acute deep vein thrombosis with or without pulmonary embolism;
11. Acute myocarditis, pericarditis or endocarditis;
12. Acute aortic dissection;
13. Intracardiac thrombus with high risk of embolism;
14. Massive pericardial effusion;
15. Those who fail to exercise adequately or refuse to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Dosage of anti-anxiety/depression drugs | Baseline and after 12 weeks of intervention
  The proportion of patients with cardiovascular diseases complicated with anxiety and depression who received a 50% reduction in the dosage of anti-anxiety/depression drugs

SECONDARY OUTCOMES:
Hamilton Depression and Anxiety Scale (HAMD, HAMA) | Baseline and at the end of the intervention (Week 12), 1 month, 6 months, 1 year and 2 years after the end of the intervention
  HAMD：0-76 points; HAMA: 0-56 points The higher the score is, the worse the result will be
Perceived Stress Scale (PSS) | Baseline and at the end of the intervention (Week 12), 1 month, 6 months, 1 year and 2 years after the end of the intervention
  PSS: 0-40 points The higher the score is, the worse the result will be
Pittsburgh Sleep Quality Index (PSQI) | Baseline and at the end of the intervention (Week 12), 1 month, 6 months, 1 year and 2 years after the end of the intervention
  PSQI: 0-21 points the higher the score, the worse the result.
12-Item Short Form Health Survey（SF-12） | Baseline and at the end of the intervention (Week 12), 1 month, 6 months, 1 year and 2 years after the end of the intervention
  SF-12:0-100 points. The higher the score, the better the health condition
Discontinuation Emergent Symptoms and Signs Scale（DESS） | Baseline and at the end of the intervention (Week 12), 1 month, 6 months, 1 year and 2 years after the end of the intervention
  The more new symptoms emerge, the more severe the adverse reactions of drug withdrawal will be.
Cardiopulmonary exercise test（CPET） | Baseline and at the end of the intervention (Week 12), one month after the end of the intervention
The recurrence rate of anxiety/depression | Baseline and one month, six months, one year and two years after the intervention ended
Electrocardiogram | Baseline and at the end of the intervention (Week 12), one month after the end of the intervention
  Evaluate QTc
Blood test | Baseline and at the end of the intervention (Week 12)
  Liver function, seven items of blood lipid, two items of myocardial function, blood routine, biochemical indicators

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No